CLINICAL TRIAL: NCT02863107
Title: Young-Onset Colorectal Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: PA11-0566; NCI-2020-07462 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PA11-0566 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2016-08-08; First posted 2016-08-11 (Estimated); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Colon Adenocarcinoma; Colorectal Carcinoma; Rectal Adenocarcinoma
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (questionnaire, biospecimen collection): PATIENTS: Patients complete questionnaires over 30-50 minutes about work, family history, medical history, health habits, and experience as a cancer survivor (quality of life, well-being, concerns, types of health care, and follow-up care received). Patients also undergo collection of blood or saliva samples. Active patients, who have undergone treatment at MD Anderson Cancer Center within the past year, complete additional questionnaires at enrollment, 6 months, 12 months after treatment completion, and then every years for up to 6 years. Also, active patients who are consented to the study more than 5 years from surgery, they may complete the survivorship questionnaire once. Patients medical records are also reviewed.
  FAMILY MEMBERS: Participants complete questionnaires over 10-15 minutes. Participants also undergo collection of blood or saliva samples once.
  Interventions: Procedure: Biospecimen Collection; Other: Medical Chart Review; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood or saliva samples
Other: Medical Chart Review — Review of medical charts
  Other Names: Chart Review
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Complete questionnaires

SUMMARY:
This study investigates the genetic factors that may influence the risk of developing colorectal cancer at a young age. Finding genetic markers for colorectal may help identify patients who are at risk of colorectal cancer. Studying individuals and families at high risk of cancer may help identify cancer genes and other persons at risk.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To define the clinical phenotype of young-onset versus (vs.) later onset colorectal cancer (CRC), including clinicopathologic characteristics, tumor molecular markers, family history, and associated lifestyle/environmental factors.

II. To examine germline genetic alterations in patients with young-onset (diagnosed between age 18 and 50), CRC and those of their first-degree relatives, in comparison to those in patients with later-onset (diagnosed at age 51 or older) CRC.

III. To determine the frequency of the mutations and pattern of inheritance of the mutations identified above in this patient population.

IV. To correlate molecular findings to clinical endpoints of survival and disease recurrence and/or progression in patients with young-onset vs. later-onset CRC.

V. To compare the treatments received by patients with young-onset vs. later-onset CRC and their subsequent survivorship experiences.

OUTLINE:

PATIENTS: Patients complete questionnaires over 30-50 minutes about work, family history, medical history, health habits, and experience as a cancer survivor (quality of life, well-being, concerns, types of health care, and follow-up care received). Active patients, who have undergone treatment at MD Anderson Cancer Center within the past year, complete additional questionnaires at enrollment, 6 months, 12 months after treatment completion, and then every years for up to 6 years. Also, active patients who are consented to the study more than 5 years from surgery, they may complete the survivorship questionnaire once. Patients medical records are also reviewed.

FAMILY MEMBERS: Participants complete questionnaires over 10-15 minutes. Participants also undergo collection of blood or saliva samples once.

ELIGIBILITY:
Inclusion Criteria:

* PATIENTS: MDACC patients who have adenocarcinoma of the colon or rectum, diagnosed between ages 18 through 50 (young-onset), or diagnosed at age 51 through 80 (later-onset)
* PATIENTS: Patient must have sufficient command of the English language and mental capacity to provide consent
* FAMILY MEMBERS: Be a parent, sibling or child (first degree blood relative) of a registered MDACC patient meeting eligibility criteria above
* FAMILY MEMBERS: Have sufficient command of the English language and mental capacity to provide consent
* FAMILY MEMBERS: Family member must be at least 18 years of age at the time of study registration

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: MD Anderson Cancer Center (MDACC) patients who have adenocarcinoma of the colon or rectum, diagnosed between ages 18 through 50 (young-onset), or diagnosed at age 51 through 80 (later-onset) and their family members
Sampling Method: Non-Probability Sample
Enrollment: 818 (Actual)
Dates: Start 2012-06-07 (Actual); Primary Completion 2030-08-31 (Estimated); Study Completion 2030-08-31 (Estimated)

PRIMARY OUTCOMES:
Clinical and epidemiologic data obtained from medical records | Up to 5 years
  Including age of colorectal cancer (CRC) diagnosis, gender, race/ethnicity, insurance status, tumor-related variables including location of the CRC, clinical and pathologic stage of CRC, histologic features including histologic grade of differentiation, mucinous histology, signet ring, and adverse features such as lymphovasucalar invasion and perineural invasion, as well as information provided from patients regarding their family history and their dietary, environmental and lifestyle information will be described using descriptive statistics. All continuous variables were described as median and interquartile range, and categorical variables as number and percentage. Comparisons between the young and the older cohorts were performed by using the Wilcoxon rank-sum test for continuous variables and Chi-squared or Fisher's exact tests for categorical variables as appropriate.
Identify polymorphism variants and/or new mutations | Up to 5 years
  Will use bioinformatic analysis to analyze and understand the identified polymorphism variants and/or new mutations. Chi-squared test will be used to test for differences between the young-onset versus (vs.) later-onset cohorts for each polymorphism variant or mutation genotype, with odds ratio and 95% confidence intervals as estimates of relative risk. A tree-based statistical approach using classification and regression tree analysis segregating study versus reference cohorts will be used. Genotypes will be coded and analyzed for the additive, dominant, recessive, or codominant models.
Treatments received including surgical, systemic, and/or radiation treatments | Up to 5 years
  Will be compared between the young and the older cohorts by using the Wilcoxon rank-sum test for continuous variables and Chi-squared or Fisher's exact tests for categorical variables as appropriate.
Degree of pathologic response to neoadjuvant chemoradiation in patients who received surgical, systemic, and/or radiation treatments | Up to 5 years
  Will be compared between the young and the older cohorts by using the Wilcoxon rank-sum test for continuous variables and Chi-squared or Fisher's exact tests for categorical variables as appropriate.
Overall response | Up to 5 years
  Will be compared between the young and the older cohorts by using the Wilcoxon rank-sum test for continuous variables and Chi-squared or Fisher's exact tests for categorical variables as appropriate.
Progression free survival | Up to 3 years
  Will be calculated. Will use Kaplan-Meier analysis to characterize the shapes of the survival curves according to normal or variant genotypes and Cox proportional hazards modeling to evaluate the association of variant genotypes, allowing for covariates such as age and stage that may vary according to genotypes and need to be controlled for evaluate evidence for an independent effect of genotype on survival or time to relapse.
Overall survival | Up to 5 years
  Will be calculated. Will use Kaplan-Meier analysis to characterize the shapes of the survival curves according to normal or variant genotypes and Cox proportional hazards modeling to evaluate the association of variant genotypes, allowing for covariates such as age and stage that may vary according to genotypes and need to be controlled for evaluate evidence for an independent effect of genotype on survival or time to relapse.
Quality of Life in Adult Cancer Survivors (QLACS) scores | Up to 5 years
  Standard scoring menu for the QLACS will be followed to obtain domain and overall scores for the QLACS. Scores will be compared between the young and older cohorts using Wilcoxon rank sum test, and the p-values will be adjusted for multiple comparisons. Mixed effects models will be constructed to analyze changes over time. In secondary analyses, quality of life scores will be stratified by disease stage, site and status. Responder bias will be assessed by comparing responders vs. non-responders for patient-, disease-, and treatment-related factors.
Adherence score | Up to 5 years
  For the survivorship care questionnaire, a summation "adherence score" will be calculated for each patient in terms of whether guideline recommended survivorship care was received by the patient. The "adherence scores" will be compared between the young vs. older cohorts using Wilcoxon rank sum test.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Qian N You, Principal Investigator — M.D. Anderson Cancer Center
Locations (5):
- United States (5):
  - MD Anderson in The Woodlands, Conroe, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - MD Anderson West Houston, Houston, Texas
  - MD Anderson League City, League City, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org